CLINICAL TRIAL: NCT04432168
Title: The TAPS Trial - Fetoscopic Laser Surgery for Twin Anemia-Polycythemia Sequence - a Multicenter Open-Label Randomized Controlled Trial
Brief Title: The TAPS Trial - Fetoscopic Laser Surgery for Twin Anemia Polycythemia Sequence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, DickOepkes, Prof. dr. D. Oepkes, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL6442700018
Record Dates: First submitted 2020-05-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Twin Anemia Polycythemia Sequence
Keywords: Monochorionic Twins; Twin-Twin Transfusion Syndrome; Fetoscopic Laser Surgery; Intrauterine Transfusion; Partial Exchange Transfusion
MeSH Terms: conditions — Fetofetal Transfusion | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fetoscopic Laser Surgery (Experimental): fetoscopic laser coagulation of the vascular anastomoses at the placental surface
  Interventions: Procedure: Fetoscopic Laser Surgery
- Standard Treatment (Other): Expectant management, IUT (with or without PET), preterm delivery
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Procedure: Fetoscopic Laser Surgery — Fetoscopic Photocoagulation of the connecting vascular anastomoses on the surface of the placenta.
  Other Names: Fetoscopic Laser Coagulation; Laser therapy; Fetoscopic Laser Ablation
  Arms: Fetoscopic Laser Surgery
Other: Standard Treatment — In the control group, the choices of treatment include expectant management, intrauterine transfusion (IUT) (with or without partial exchange transfusion (PET)) or preterm delivery, depending on the judgment of the fetal surgeon with regard to the gestational age and state of the disease.
  * Expectant management will consist of close monitoring with ultrasound including Doppler measurements of the middle cerebral artery peak systolic velocity (MCA-PSV), at least every week.
  * IUT: the intrauterine infusion of red blood cells into the circulation of the donor twin treat anemia.
  * PET: the intrauterine infusion of saline into the circulation of the recipient twin to treat polycythemia.
  * Preterm delivery: Induction of labor or cesarean section before 36 weeks of gestation.
  Arms: Standard Treatment

SUMMARY:
This multicenter open-label randomized controlled trial is set up to evaluate the effect of fetoscopic laser surgery on the gestational age at birth for monochorionic twin pregnancies diagnosed with twin anemia-polycythemia sequence. Half op the patients will be treated with fetoscopic laser surgery, while the other half will be managed with standard treatment. The hypothesis is that fetoscopic laser therapy will improve neonatal outcome by prolonging pregnancy.

DETAILED DESCRIPTION:
Rationale: Monochorionic twins share one placenta and are connected to each other via vascular anastomoses at the placental surface, allowing the blood to transfer bi-directionally between the two fetuses. Unbalanced inter-twin blood transfusion can result in twin anemia-polycythemia sequence (TAPS). Management options include: fetoscopic laser surgery, intrauterine blood transfusion (IUT) with or without partial exchange transfusion (PET), preterm delivery, selective feticide and expectant management. The optimal treatment for TAPS is not clear. Fetoscopic laser surgery is the only causative treatment option, but data on the feasibility of this procedure are mainly based on case reports and small cohort studies. A large randomized controlled trial is needed to evaluate the possible beneficial effect of fetoscopic laser surgery and to determine the optimal treatment option for TAPS.

Objective: The aim of this trial is to investigate whether fetoscopic laser surgery improves the outcome for TAPS twins as compared to the control group (standard care consisting of expectant management, IUT, preterm delivery). The hypothesis is that fetoscopic laser therapy will improve neonatal outcome by prolonging pregnancy.

Study design: International multi-centered open-label randomized controlled trial to assess whether fetoscopic laser surgery (experimental group) improves the outcome of TAPS twins compared to standard care (control group).

Study population: Monochorionic twin pregnancies with TAPS stage ≥ 2 (spontaneous or post-laser) diagnosed between 20 and 28 weeks of gestation.

Intervention: In the experimental group fetoscopic laser surgery is performed, whereas the control group is treated with standard care (expectant management, IUT (with PET), selective feticide and/or preterm delivery, depending on the opinion of the fetal surgeon).

Main study endpoints: The primary outcome is gestational age at birth. Secondary outcomes include: perinatal mortality or severe neonatal morbidity, hematological complication, procedure related complications and long-term neurodevelopmental outcome at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Monochorionic twin pregnancy complicated by either spontaneous or post-laser twin anemia polycythemia sequence (TAPS), stage ≥ 2, diagnosed between 20+0 and till 28+0 weeks of gestation
* Women aged 18 years or more, who are able to consent.
* Written informed consent to participate in this randomized controlled trial, forms being approved by the Ethical Committees.

Exclusion Criteria:

* TAPS stage 1
* TAPS stage≥ 2, diagnosed within 1 week after laser surgery for twin-twin transfusion syndrome (TTTS) (a large inter-twin middle cerebral artery peak systolic velocity difference within a week after laser for TTTS is likely to related to hemodynamic reequilibration, and is usually not based on TAPS)
* Triplet pregnancies, or higher order multiple pregnancies
* TAPS cases that already underwent an intrauterine treatment (with the exception of laser surgery for TTTS in post-laser TAPS cases)
* Congenital abnormalities (including severe cerebral injury) in one or both twins

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Gestational Age at Birth | 2 weeks after expected date of birth
  Gestational age: completed weeks + additional days since the first day of the last menstruational period of the mother.

SECONDARY OUTCOMES:
Number of patients with perinatal mortality | 42 days (28 days neonatal period+2 weeks postdates) after expected date of birth
  Perinatal mortality is defined as fetal death or neonatal death (demise of a liveborn child within 28 days after birth)
Number of patients with severe neonatal morbidity | 42 days (28 days neonatal period+2 weeks postdates) after expected date of birth
  Severe neonatal morbidity is defined as the presence of at least one of the following:
  * Respiratory distress syndrome requiring surfactant or mechanical ventilation
  * Proven early onset neonatal sepsis with positive blood cultures within 72 hours postpartum
  * Retinopathy of prematurity stage 3 or higher
  * Necrotizing enterocolitis stage 2 or higher
  * Patent ductus arteriosus requiring medical therapy or surgical closure
  * Severe cerebral injury (defined as intraventricular hemorrhage grade 3 or higher, cystic periventricular leukomalacia grade 2 or higher, ventricular dilatation greater than the 97th centile, porencephalic or parenchymal cysts or other severe cerebral lesions)
Number of patients with hematological complications | 2 weeks after expected date of birth
  Hematological complications are defined as the presence of at least one of the following:
  * Anemia in donor requiring a blood transfusion within 24 hours after birth
  * Polycythemia in recipient requiring a partial exchange transfusion within 24 hours after birth
  * necrotic skin injury
  * limb ischemia
  * platelet count < 150,000/microL
  * albumin levels < 20 g/L
  * protein levels < 40 g/L
Number of patients with procedure-related complications | 2 weeks after expected date of birth
  Procedure-related complications are defined as at least one of the following:
  * amniotic band syndrome
  * iatrogenic monoamnionicity
  * Preterm premature rupture of the membranes
  * Placental abruption
  * clinical chorioamnionitis
  * histological chorioamnionitis and/or funisitis
Number of patient with mild neurodevelopmental impairment | 2 years after expected date of birth
  Mild neurodevelopmental impairment is defined as at least one of the following:
  * cerebral palsy (spastic bilateral, spastic unilateral, or mixed)
  * Impaired cognitive or motor development defined as Score < 85 (1 standard deviation (SD) below the mean) as assessed by Bayley Scales of Infant and Toddler Development version 3 (BSID-III)
  * Impaired functioning in communication, fine and gross motor, problem solving, personal and social functioning defined as Score > 1 SD below the mean as assessed by Ages and Stages Questionnaire version 3 (ASQ-III)
  * severe visual loss (blind or partially sighted)
  * severe hearing loss (needing hearing aids)
Number of patients with severe neurodevelopmental impairment | 2 years after expected date of birth
  Severe neurodevelopmental impairment is defined as at least one of the following:
  * cerebral palsy defined as a gross motor function classification system (CMFCS) grade > 1
  * Impaired cognitive or motor development defined as a score < 70 (2 SD below the mean) as assessed by the Bayley Scales of Infant and Toddler Development version 3 (BSID-III)
  * Impaired functioning in communication, fine and gross motor, problem solving, personal and social functioning defined as a score > 2 SD below the mean as assessed by Ages and Stages Questionnaire version 3 (ASQ-III)
  * Bilateral blindness defined as visual acuity of less than 3/60 in the better eye
  * Bilateral deafness defined as severe or profound hearing loss in both ears (severe hearing loss: a person can only hear sounds > 70-89 decibel , profound hearing loss: a person can only hear sounds > 90 decibel
Number of patients with behavioral problems | 2 years after expected date of birth
  Behavioral problems are defined as a T-score ≥ 64 for one of the following broad band scales: total problem score, Internalizing problems (anxious/depressed, withdrawn, somatic complaints), Externalizing problems (rule-breaking, aggressive behavior) as measured with the Child Behaviour Checklist 1.5-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dick Oepkes, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (5):
- Yale University, New Haven, Connecticut, United States
- Vittore Buzzi Children's Hospital, Milan, Lombardy, Italy
- Leiden University Medical Center, Leiden, South Holland, Netherlands
- Vall d'Hebron University Hospital, Barcelona, Spain
- Karolinska University Hospital, Stockholm, Södermanland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopriore E, Middeldorp JM, Oepkes D, Kanhai HH, Walther FJ, Vandenbussche FP. Twin anemia-polycythemia sequence in two monochorionic twin pairs without oligo-polyhydramnios sequence. Placenta. 2007 Jan;28(1):47-51. doi: 10.1016/j.placenta.2006.01.010. Epub 2006 Mar 3. PMID 16516289
- [Background] Robyr R, Lewi L, Salomon LJ, Yamamoto M, Bernard JP, Deprest J, Ville Y. Prevalence and management of late fetal complications following successful selective laser coagulation of chorionic plate anastomoses in twin-to-twin transfusion syndrome. Am J Obstet Gynecol. 2006 Mar;194(3):796-803. doi: 10.1016/j.ajog.2005.08.069. PMID 16522415
- [Background] Sananes N, Veujoz M, Severac F, Barthoulot M, Meyer N, Weingertner AS, Kohler M, Guerra F, Gaudineau A, Nisand I, Favre R. Evaluation of the Utility of in utero Treatment of Twin Anemia-Polycythemia Sequence. Fetal Diagn Ther. 2015;38(3):170-8. doi: 10.1159/000380822. Epub 2015 Mar 17. PMID 25790745
- [Background] Slaghekke F, Favre R, Peeters SH, Middeldorp JM, Weingertner AS, van Zwet EW, Klumper FJ, Oepkes D, Lopriore E. Laser surgery as a management option for twin anemia-polycythemia sequence. Ultrasound Obstet Gynecol. 2014 Sep;44(3):304-10. doi: 10.1002/uog.13382. Epub 2014 Aug 4. PMID 24706478